CLINICAL TRIAL: NCT05632692
Title: Menthol Mouth Rinsing and Performance Responses of Elite Football Referees in the Heat: a Randomized Crossover Trial
Brief Title: Menthol Mouth Rinsing and Performance Responses of Elite Football Referees in the Heat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 20/2021/CEFCNAUP/2021
Record Dates: First submitted 2022-11-08; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-10

CONDITIONS: Exercise Induced Hyperthermia; Performance Demands of Exercising in the Heat

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A menthol solution is going to be formulated by crushing and dissolving one noncalorific menthol candy drop (15 mg) in 150 ml of warm water, in order to obtain a solution with a concentration of 0.01%. Prior to use, solutions are going to be aliquoted for mouth rinse and warmed at room temperature. Then, it will be served to each participant on individual bottles in a total dose of 75 ml before exercise and 75 ml during exercise.
  Interventions: Other: Menthol solution
- Placebo (Placebo Comparator): A placebo beverage is going to be prepared using noncaloric berry-flavored sweetener consisting of sucralose candy drops, which will be crushed and dissolved in 150 ml of warm water. Prior to use, solutions are going to be aliquoted for mouth rinse and warmed at room temperature. Then, it will be served to each athlete on individual bottles in a total dose of 75 ml before exercise and 75 ml during exercise.
  Interventions: Other: Menthol solution

INTERVENTIONS:
Other: Menthol solution — Menthol application, through oral solutions, stimulates the mandibular and maxillary branches of the trigeminal nerve (which are predominantly responsible for detection of temperature and nociceptive stimuli across the face and within the oral cavity) and has consistently shown to improve thermal comfort and decrease thermal sensation, which are thought to modulate perceived exertion to improve performance in the heat.

SUMMARY:
Ten male football referees will be recruited to perform two intermittent football protocols , separated by at least 7 days (wash-out period). After passing the eligibility criteria, the participants will be randomly assigned, according to a computer-generated allocation schedule, to 1 of 2 beverages sequences: (1) intervention - menthol solution 0.01% (room temperature) and (2) placebo - noncaloric berry-flavoured solution (room temperature). The participants will be provided with one of the 2 beverages before warm-up (pre-cooling) and at the half-time (per-cooling). The trials will follow a randomised counterbalanced crossover design, blinded to the participants, and will take place in indoor facilities, where WBGT exceed 30◦C, at the same time of the day, to control for circadian variations. Each trial involves an exercise protocol (SAFT-90), lasting 90 minutes, separated into two 45-minute parts. The first half will be preceded by a warm-up and the second half by a 15-minute break.

The results of this study are expected to determine whether mouth rinsing a menthol solution, before a football exercise protocol performed in the heat, will help to alleviate physiological strain and improve performance parameters, comparing to a non-cooling strategy, in elite male football referees. Thus, we can be closer to defining nutritional strategies of internal cooling, that will be an advantage for the performance of the football referees, concretely in the competitions carried out under adverse environmental conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male football referees aged over 18 and under 45 years;
2. With normal weight (BMI ≥ 18.5 and ≤ 24.9 kg/m2);
3. Availability to participate in the introductory meeting, familiarization session and 2 experimental sessions;
4. Ability to read and sign the informed consent.

Exclusion Criteria:

1. Under the influence of any medications that may affect urinary parameters, thermoregulation mechanisms, circulatory system, thyroid and pituitary function or metabolic status;
2. Injury, diabetes, autoimmune disease, cardiovascular disease or obstructive disease of the gastrointestinal tract (e.g., diverticulitis, inflammatory bowel disease);
3. Schizophrenia, bipolar disorder or other psychotic disorders;
4. Eating disorders;
5. MRI scans scheduled within 48 hours after familiarization session or any of the experimental trials.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate change | A change in heart rate from baseline (immediately before exercise) to each 15-minute block of the exercise protocol will be assessed.
  Heart rate is a physiological parameter of performance and will be measured through HR monitors (Polar H10 Heart Rate Sensor, USA). PolarH10 can accurately measure mean HR and low-frequency oscillations (up to 0.15 Hz) of HR at rest and during exercise.
Sweating rate at the first half | Sweating rate is going to be calculated at the end of the first half of the exercise protocol (after 45 min of exercise)
  Sweating rate is a physiological parameter of performance and is going to be calculated recurring to the following equation : SR= (Pre exercise body weight - postexercise body weight + fluid intake - urine volume)/(exercise time in hours).
Sweating rate at the second half | Sweating rate is going to be calculated at the end of the second half of the exercise protocol (after 90 min of exercise)
  Sweating rate is a physiological parameter of performance and is going to be calculated recurring to the following equation : SR= (Pre exercise body weight - postexercise body weight + fluid intake - urine volume)/(exercise time in hours).
Core temperature change | A change in core temperature from baseline (immediately before exercise) to each 15-minute block of the exercise protocol will be assessed
  Core temperature is a physiological parameter of performance and can be accessed using a telemetric pill ingested 30 minutes prior the start of the exercise (BodyCap®, France). Due to the good measuring accuracy, the ability to measure in field-based situations and the non-invasive character of this temperature measurement method, the ingestible telemetric temperature pill is suitable to assess core temperature during exercise
Ratings of perceived exertion (RPE) | RPE is going to be accessed at the end of the exercise protocol.
  RPE is a subjective psychological/perceptual parameter that impacts performance and will be recorded through CR-10 Borg scale that goes from 0 ("rest") to 10 ("maximal effort").
Thermal comfort (TC) change | A change in TC from baseline (immediately before intervention) to after intervention and to each 15-minute block of the exercise protocol will be assessed.
  TC is a subjective psychological/perceptual parameter that influences performance and is going to be accessed according to a 6-point scale from to -3 ("very uncomfortable) to 3 ("very comfortable").
Thermal sensation (TS) change | A change in TS from baseline (immediately before intervention) to after intervention and to each 15-minute block of the exercise protocol will be assessed.
  TS is a subjective psychological/perceptual parameter that impacts performance and will be recorded with a 9-point scale from -4 ("very cold") to 4 ("very warm").
Perceived thirst (PT) change | A change in PT from baseline (immediately before intervention) to after intervention and to each 15-minute block of the exercise protocol will be assessed.
  PT is a subjective marker of hydration status and will be evaluated recurring to a 7-point scale from 1 ("not thirsty at all") to 7 ("very, very thirsty")
Physical performance change | A change in each physical performance indicator from baseline (immediately after the warm-up) to each 15-minute block of the exercise protocol will be assessed
  Physical performance responses will be measured using 100 Hz accelerometery, with Sonda 4.0 software (StatSports®, UK) to estimate total distance, sprint distance, accelerations and decelerations number

SECONDARY OUTCOMES:
Hydration status before | Hydration status is going to be recorder at baseline (pre-exercise)
  Hydration status is going to be assessed recurring to urine test strip (Combur10 Test M, Roche) and Urisys 1100® analyser (Roche, Switzerland).
Hydration status after | Hydration status is going to be recorder at the end of the exercise protocol
  Hydration status is going to be assessed recurring to urine test strip (Combur10 Test M, Roche) and Urisys 1100® analyser (Roche, Switzerland).
Ad libitum fluid intake at the first half | Ad libitum fluid intake is going to be assessed at the end of the first half of the exercise protocol (after 45 min of exercise)
  Fluid intake is going to be recorded via the measurement of mass change of the individual bottles provided to the referees at the warm-up and at the end of the session, to the nearest 0.1 ml (Seca, Hamburg, Germany).
Ad libitum fluid intake at the second half | Ad libitum fluid intake is going to be assessed at the end of the second half of the exercise protocol (after 90 min of exercise)
  Fluid intake is going to be recorded via the measurement of mass change of the individual bottles provided to the referees at the warm-up and at the end of the session, to the nearest 0.1 ml (Seca, Hamburg, Germany).
Blood lactate levels before | Blood lactate levels are going to be recorded before the start of the exercise protocol
  Blood lactate levels will be measured recurring to a Blood Lactate Meter (Lactate Pro 2, Arkray, U.S.A).
Blood glucose levels before | Blood glucose levels are going to be recorded before the start of the exercise protocol
  Blood glucose levels will be measured recurring to a Glucometer (FreeStyle Precision Neo, Abbott Laboratories, U.S.A).
Blood glucose levels after | Blood glucose levels are going to be recorded immediately after the end of the exercise protocol
  Blood glucose levels will be measured recurring to a Glucometer (FreeStyle Precision Neo, Abbott Laboratories, U.S.A).
Blood lactate levels after | Blood lactate levels are going to be recorded immediately after the end of the exercise protocol
  Blood lactate levels will be measured recurring to a Blood Lactate Meter (Lactate Pro 2, Arkray, U.S.A).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roriz M, Brito J, Teixeira FJ, Spyrou K, Teixeira VH. The effect of menthol rinsing before intermittent exercise on physiological, physical, and thermo-behavioral responses of male football referees in hot and humid environment. Front Sports Act Living. 2024 Jan 22;6:1334739. doi: 10.3389/fspor.2024.1334739. eCollection 2024. PMID 38318484
- [Derived] Roriz M, Brito J, Teixeira FJ, Spyrou K, Teixeira VH. Menthol mouth rinsing and performance in elite football referees in the heat: A study protocol for a randomized crossover trial. Contemp Clin Trials Commun. 2023 Aug 22;35:101202. doi: 10.1016/j.conctc.2023.101202. eCollection 2023 Oct. PMID 37691850